CLINICAL TRIAL: NCT04884152
Title: Investigation of the Effectiveness of Telerehabilitation in Individuals Myofascial Temporomandibular Dysfunction With Bruxism
Brief Title: Telerehabilitation in Individuals Temporomandibular Dysfunction With Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Ezgi Hatice Giray, Research assistant, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/012
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2022-08

CONDITIONS: Myofascial Pain; Temporomandibular Disorder; Bruxism
Keywords: Myofascial Pain; Temporomandibular Disorder; Bruxism; Telerehabilitation
MeSH Terms: conditions — Temporomandibular Joint Disorders; Bruxism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Exercise Group (Active Comparator): The home Exercise program includes an educational training program about parafunctional activities of patients having bruxism with myofascial temporomandibular disorders. The program includes stretching and strengthening of masticatory and neck muscles and posture exercises as well as diaphragmatic breathing exercises.
  Relaxation: Relaxation exercises with diaphragmatic breathing Posture Exercise: Rest position of tongue and TMJ, head and neck posture correction exercises Stretching Exercises: Stretching exercises for chewing muscles, cervical muscles, and pectoral muscles Strengthening: The neck will consist of strengthening exercises for deep flexor muscles, suprahyoid and infrahyoid muscles, and scapular retractors.
  Interventions: Procedure: Home Exercise Group
- Telerehabilitation Group (Experimental): The program includes the same stretching and strengthening of masticatory and neck muscles and posture exercises as well as diaphragmatic breathing exercises using telerehabilitation once a week by video call, and reminder messages will be sent to the patients 3 times a week.
  Relaxation: Relaxation exercises with diaphragmatic breathing Posture Exercise: Rest position of tongue and TMJ, head and neck posture correction exercises Stretching Exercises: Stretching exercises for chewing muscles, cervical muscles, and pectoral muscles Strengthening: The neck will consist of strengthening exercises for deep flexor muscles, suprahyoid and infrahyoid muscles, and scapular retractors.
  Interventions: Procedure: Telerehabilitation Group

INTERVENTIONS:
Procedure: Home Exercise Group — Educational training program about bruxism and the other oral parafunctional activities in patients with myofascial temporomandibular disorders.
  Arms: Home Exercise Group
Procedure: Telerehabilitation Group — Telerehabilitation program combined with educational training program about bruxism and the other oral parafunctional activities in patients with myofascial temporomandibular disorders.
  Arms: Telerehabilitation Group

SUMMARY:
The aim of the study is to compare the effects of Home Exercise Therapy (HET) and Telerehabilitation in patients with myofascial temporomandibular disorders (TMD)with bruxism.

DETAILED DESCRIPTION:
Home Exercise will be Group 1 and Telerehabilitation group will be Group 2.

Group 1 HET, will include an educational training program about parafunctional activities of TMD disorders and bruxism and active exercises for 4 weeks.

As part of the Home exercise program, a written document will be prepared, including relaxation, breathing training, posture, stretching, and strengthening exercises to be given to the patients.

Group 2, in addition to the training and written document, the second group will receive the same exercises using telerehabilitation once a week by video call, and reminder messages will be sent to the patients 3 times a week.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 65 years old
* Patients with TMD in the myofascial Group Ia, Ib according to the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) and diagnosed with bruxism
* Having pain ≥ 3 according to the Visual Analog Scale
* Those who have not received medical treatment for the last 3 months and will not receive it during the treatment process will be included in the study.

Exclusion Criteria:

* Ages under 18 and over 65 years old
* Patients with disc displacement and/or TMJ degeneration
* Patients who have orthodontic or splint treatment
* Patients with musculoskeletal problems in which systemic specific pathological conditions such as cervical and/or temporomandibular joint (TMJ) problem malignancy, fracture, the rheumatoid disease is proven
* Patients who have undergone any surgery related to the cervical and/or TMJ
* Patients with facial paralysis
* Patients who regularly use analgesic or anti-inflammatory drugs
* Patients who have received physical therapy associated with TMJ in less than 3 months
* Patients with a history of trauma (whiplash injury, condylar trauma, fracture)
* Patients with cognitive deficits
* Participation rate lower than 80% of the program schedule

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain at 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
  Visual Analog Scale will be used where patients will be asked to rate their pain on a scale from 0 to 10 with 0 indicating no pain and 10 the maximum worst pain, at the baseline and the end of 4 weeks intervention and at the end 8 weeks from baseline.
Change from Baseline in Mandibular range of movements at 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
  Maximum mouth opening, mandibular lateral right and left shift, and mandibular protrusion range of motion measurements in mm.
Change from Baseline in Neck disability at 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
  Neck Disability Index, consisting of a total of ten titles, was developed by Vernon and Mior in 1991. It includes topics such as pain intensity in the neck, personal care, lifting, reading, headaches, concentration, driving, sleep, and leisure activities. The maximum score is 50, while the minimum is 0 points.
  Classification according to total score is as follows: 0-4 (no restrictions); 5-14 (mild restriction); 15-24 (moderate restriction); 25-34 (severe limitation); 34 and above (completely limited).
Change from Baseline in Headache at 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
  Headache Impact Test-6 test consists of 6 questions about the severity of headache, the effect of pain on daily life activities, how often it causes fatigue and low motivation, and concentration impairment. Scoring is done between 36-78.
Change from Baseline in Sleep Quality at 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
  Pittsburg Sleep Quality Index test is used to evaluate sleep effects in the last few months. This questionnaire contains 24 questions, 19 of which are personal, and 5 of which are to be answered by a partner about sleep during both day and night. Five questions answered by the partner are not included in the scoring. Self-assessment questions contain different items related to sleep quality, which provide information about sleep duration, latency, and the frequency and severity of specific sleep problems. The total score is between 0-21. A score of 5 and below indicates good sleep quality, and a score above 5 indicates poor sleep quality.
Change from Baseline in Oral Behavior at 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
  Evaluation of oral habits with the Oral Habits Questionnaire consisting of 21 items, each item was evaluated according to the frequency of complaints as "4 = always; 3 = most of the time; 2 = sometimes; 1 = several times or 0 = none". The questions cover the times of sleep and wakefulness. The overall score ranges from 0 to 84.
Change from Baseline in Quality of life at 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
  The individual's personal perception of how oral health affects their quality of life and general health is measured. Oral Health Impact Profile-14 is a scale system that evaluates this perception with questions for functional limitation, physical pain, psychological discomfort, physical, psychological and social inadequacy, and disability measures. It is concluded that as the total score increases, the severity of the problem increases, and the quality of life decreases.

SECONDARY OUTCOMES:
Change from Baseline in Head and Shoulder Posture at 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
  Forward Head Posture: The angle between the C7-Ear-Horizontal plane in the sitting position (in degrees with a goniometer) Shoulder Posture: The angle between the Acromion-C7-Horizontal Plane in the sitting position (in degrees with a goniometer).
Change from Baseline in Anxiety at 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
  The State-Trait Anxiety Inventory was developed by Spielberger et al. to measure state anxiety and trait anxiety. The questionnaire consists of 40 questions, the expressions used by the person in expressing his own feelings were included. There are four categories (nothing-a little-much-completely) for answers.
Change from Baseline in Fatigue at 4 weeks and 8 weeks | Baseline, 4 weeks, 8 weeks
  The Fatigue Severity Scale is used to measure the severity of fatigue in the past week, including today. The questionnaire consists of 9 items in total, and participants are asked to give a score from 1 to 7 for each question. The fatigue level of the patient is determined according to the score obtained by the sum of the points. The higher the level of fatigue, the higher the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, Study Director — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)